CLINICAL TRIAL: NCT01592890
Title: Single-centre, Open-label Study Investigating the Excretion Balance, Pharmacokinetics and Metabolism of a Single Dose of 14C-labeled RO4917523 and an Intravenous Tracer Dose of 13C-labeled RO4917523 in Healthy Male Volunteers
Brief Title: A Study of The Excretion Balance, Pharmacokinetics and Metabolism of A Single Oral Dose of [14C]-Labeled RO4917523 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: BP27854; 2011-004597-28 (EudraCT Number)
Record Dates: First submitted 2012-05-04; First posted 2012-05-07 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

ARMS (1):
- [14C]-labeled RO4917523 (Experimental)
  Interventions: Drug: RO4917523

INTERVENTIONS:
Drug: RO4917523 — [14C]-labeled RO4917523, single oral dose
Drug: RO4917523 — [13C]-labeled RO4917523, single intravenous tracer dose

SUMMARY:
This single-center, open-label study will assess the excretion balance, pharmacokinetics and metabolism of oral [14C]-labeled RO4917523 in healthy male volunteers. Subjects will receive a single oral dose of [14C]-labeled RO4917523 and an intravenous tracer dose of [13C]-labeled RO4917523 on Day 1. In-clinic period will be up to 18 Days. Anticipated time on study is up to 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male adults, 18 to 65 years of age inclusive
* Body mass index (BMI) 18.0 to 32.0 kg/m2
* Healthy, as judged by a physician on the basis of a medical history, general physical examination, laboratory tests, vital signs and 12-lead ECG
* Medical history without major pathology
* Agree to use two effective methods of contraception with their partners, including one barrier method (e.g. condom) throughout the study and for up to 3 months after the last dose of study drug

Exclusion Criteria:

* History of relevant drug and or food allergies
* Smoking (within 60 days prior to drug administration until the follow-up visit)
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products)
* Participation in a drug study within 60 days preceding first administration of study drug; participation in more than 3 other drug studies within 10 months preceding the first administration of study drug
* Infrequent bowel movements (less than once per 2 days)
* Participation in another ADME study with a radiation burden >0,1 mSv in the period of 1 years before the start of the study
* Positive screen for drugs of abuse
* Average intake of more than 24 units of alcohol per week
* Positive for hepatitis B, hepatitis C or HIV infection

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Elimination: urinary and fecal recovery of total radioactivity | Pre-dose and up to approximately Day 18 post-dose
Plasma concentrations of RO4917523 | Pre-dose and up to approximately Day 18 post-dose

SECONDARY OUTCOMES:
Metabolites of RO4917523 in plasma/urine/blood pellet/feces based on radioactive metabolic profiling | Pre-dose and up to approximately Day 18 post-dose
Absolute bioavailability: Area under the concentration-time curve (AUC) | Pre-dose and up to approximately Day 18 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Zuidlaren, Netherlands